CLINICAL TRIAL: NCT05004688
Title: An Open-label Trial to Evaluate the Effects of BCG Immunization on Biomarkers of Inflammation/Immune Response and Alzheimer's Disease in Adults With Mild Cognitive Impairment and Mild-to-Moderate Dementia Due to Alzheimer's Disease
Brief Title: A Trial to Evaluate the Effects of BCG in Adults With MCI and Mild-to-Moderate AD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Steven E Arnold, MD (Other)
Responsible Party: Sponsor-Investigator, Steven E Arnold, MD, Professor of Neurology, Massachusetts General Hospital
Organization: Massachusetts General Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2021P002577
Record Dates: First submitted 2021-08-06; First posted 2021-08-13 (Actual); Results first posted 2025-04-13 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-03

CONDITIONS: Mild Cognitive Impairment; Mild Dementia; Moderate Dementia; Alzheimer Disease
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease | interventions — Biological Products; BCG Vaccine

STUDY DESIGN:
Intervention Model Description: open-label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- BCG (Experimental): Active BCG immunization
  Interventions: Biological: Biological/Vaccine: Bacillus Calmette-Guerin (BCG)

INTERVENTIONS:
Biological: Biological/Vaccine: Bacillus Calmette-Guerin (BCG) — Two Bacillus Calmette-Guérin (Japan BCG) vaccine injections spaced four week apart. Each injection will have 0.36-3.9 x 10^6 colony forming units (CFU) reconstituted in 0.1 mL saline.
  Other Names: BCG

SUMMARY:
A study of the effects of Bacillus Calmette-Guérin (BCG) immunization on cerebrospinal fluid and blood-based biomarkers in older with mild cognitive impairment and mild-to-moderate to Alzheimer's disease.

DETAILED DESCRIPTION:
This single-site, open-label trial will investigate the effects of BCG vaccination on IIR and AD biofluid biomarkers, magnetic resonance imaging (MRI) biomarkers, and neurocognitive/behavioral functioning over a one year period in older adults with mild cognitive impairment (MCI) to mild-to-moderate dementia due to AD. This study will also gather data on tolerability and safety.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals between the ages of 55-85;
2. MCI or moderate dementia due to AD as defined by the 2011 NIA-AA Workgroup recommendations;
3. MoCA ≥ 8 at screening;
4. Global CDR between 0.5-2 (inclusive) at screening;
5. Amyloid and/or tau biomarkers indicative of AD pathology;
6. Education level, English language skills and literacy indicates subject will be able to complete all assessments;
7. Has a study partner who, in the investigator's judgement, has frequent, direct contact with the participant at least several days a week, can accompany the participant to all visits, and is also able to provide information to study investigator/staff;
8. Willing and able to complete all assessment and study procedures, including blood and lumbar punctures, and clinical assessments;
9. If on cholinesterase inhibitor and/or memantine, doses are stable for 3 months prior to baseline;
10. Negative test results for HIV antibody and Tuberculosis (QuantiFERON) at screening;
11. No prior BCG exposure either through birth vaccinations (born in North American) or BCG bladder cancer treatment.

Exclusion Criteria:

1. History of chronic infectious disease, such as HIV or untreated or active hepatitis;
2. History of tuberculosis, positive interferon-gamma release assay (IGRA, also known as the QuantiFERON-TB test), including a test with a high reactivity to mycobacteria of non-tuberculosis variety;
3. Prior BCG vaccination, positive T-spot tuberculosis test or a T-spot test showing significant Mycobacteria exposure;
4. A positive SARS-CoV-2 PCR result within 3 months of screening, or known close contact with a confirmed COVID-19 positive person or symptoms highly suspicious for COVID-19 (per CDC guidelines) within 1 month of screening, including fever, cough, shortness of breath, chills, muscle pain, new loss of taste or smell, vomiting or diarrhea, and/or sore throat, based on clinician's judgment;
5. History of treatment with metformin within the past one year;
6. Treatment with other investigational agents which, at the discretion of the investigator, interfere with safety and/or study outcomes;
7. Current treatment with immunosuppressants (calcineurin inhibitors, corticosteroids, or biological or cytotoxic immunosuppressants, or disease or condition likely to require high dose steroid or immunosuppressive therapy);
8. Other conditions or treatments associated with increased risk of infections or treatment with immunosuppressive medications for any reason;
9. Current treatment with aspirin > 160 mg/day or chronic, daily NSAIDs;
10. Current (as of time of study screening) or chronic use of antibiotics;
11. History of keloid formation;
12. Living with someone who is immunosuppressed and/or at high risk for infectious diseases (for example, HIV+ or taking immunosuppressive medications for any reason), or in a job (e.g. healthcare) in which the subject works with immunosuppressed populations;
13. Other/confounding neurological or psychiatric condition, unstable medical or psychiatric conditions, contraindications to BCG use and lab abnormalities or concurrent medication use posing risk for BCG or study procedures;
14. Laboratory abnormalities in B12, Folate, TSH, or other common laboratory parameters that may contribute to cognitive dysfunction per clinician judgment;
15. Laboratory abnormalities in CBC, electrolytes, LFTs, BUN, Cr, total serum immunoglobulins, ESR, CRP, or urinalysis posing risk to treatment with BCG per clinician judgment;
16. Laboratory abnormalities in PT-INR, which would pose a risk to performing the lumbar puncture procedure;
17. Discontinuation of cholinesterase inhibitor or memantine within one month (28 days) prior to baseline visit;
18. Females who are pregnant, lactating or of child-bearing potential;
19. If male with female partner(s) of childbearing potential, unwilling or unable to adhere to contraception requirements specified in the protocol.
20. Administration of live vaccine within 30 days of screening visit or BCG immunizations
21. Administration of non-live vaccine within 14 days of screening visit or BCG immunizations
22. If participating in optional MRI: Existing contraindication to MRI per MGH Athinoula A. Martinos Center research guidelines

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2022-03-25 (Actual); Primary Completion 2024-01-15 (Actual); Study Completion 2024-01-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Arnold, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Alzheimer's Clinical and Translational Research Unit, Charlestown, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Active BCG Immunization: Active BCG immunization
  Biological/Vaccine: Bacillus Calmette-Guerin (BCG): Two Bacillus Calmette-Guérin (Japan BCG) vaccine injections spaced four week apart. Each injection will have 0.36-3.9 x 10^6 colony forming units (CFU) reconstituted in 0.1 mL saline.
Period: Overall Study
Arm/Group | Active BCG Immunization
Started | 15
Completed | 4
Not Completed | 11
Not completed — Protocol Violation | 7
Not completed — Physician Decision | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Active BCG Immunization
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 15
  More than one race | 0
  Unknown or Not Reported | 0
CSF Collected [Count of Participants; unit: Participants] | 7
Blood Collected [Count of Participants; unit: Participants] | 7
Cognitive testing measured [Count of Participants; unit: Participants] | 7

OUTCOME MEASURES:

1. Primary Outcome: Blood Biomarkers of Pharmacodynamic Response- Cytokines
Description: Change in concentration (Average difference) of circulating cytokines in blood from baseline (Average difference).Cytokines include: Plasma IFN-g (pg/ml), Plasma IL-1b (pg/ml), Plasma IL-2 (pg/ml), Plasma IL-6 (pg/ml), Plasma IL-10 (pg/ml), Plasma TNF-a (pg/ml).
  Mean differences (and standard deviations) from baseline values are presented for the Day 364 (end of study) sample collections for the 4 participants in the study.
Time Frame: Baseline to Day 364
Measure: Mean (Standard Deviation); unit: picogram/milliliter (pg/ml)
Groups:
- Active BCG Immunization: Biological/Vaccine: Bacillus Calmette-Guerin (BCG): Two Bacillus Calmette-Guérin (Japan BCG) vaccine injections spaced four week apart. Each injection will have 0.36-3.9 x 10^6 colony forming units (CFU) reconstituted in 0.1 mL saline.
Arm/Group | Active BCG Immunization
Number analyzed (Participants) | 4
picogram/milliliter (pg/ml)
  Plasma IFN-g (pg/ml) | 26.672 (125.864)
  Plasma IL-1b (pg/ml) | 190.829 (181.329)
  Plasma IL-2 (pg/ml) | 20.309 (19.205)
  Plasma IL-6 (pg/ml) | 2293.879 (4308.539)
  Plasma IL-10 (pg/ml) | 366.090 (656.157)
  Plasma TNF-a (pg/ml) | 53.903 (54.002)

2. Primary Outcome: CSF Biomarkers of Pharmacodynamic Response- Cytokines
Description: Change in concentration (Average difference) of circulating cytokines in CSF from baseline (Average difference). Cytokines measured include: CSF IFN-g (pg/ml), CSF IL-1b (pg/ml), CSF IL-2 (pg/ml), CSF IL-6 (pg/ml), CSF IL-10 (pg/ml), CSF TNF-a (pg/ml).
  Mean differences (and standard deviations) from baseline values are presented for the Day 84 sample collections for the 7 participants with complete data in the study.
Time Frame: Baseline to Day 84
Population: Since this outcome was analyzing the average difference between Day 0 and Day 84, there were more participants enrolled for these times points than when comparing Day 0 to Day 364. 15 participants started the trial, and only 4 completed, thus there were 7 active participants for the Day 84 timepoint.
Measure: Mean (Standard Deviation); unit: picogram/milliliter (pg/ml)
Arm/Group | Active BCG Immunization
Number analyzed (Participants) | 7
picogram/milliliter (pg/ml)
  CSF IFN-g (pg/ml) | 0.053 (13.002)
  CSF IL-1b (pg/ml) | -1.287 (15.192)
  CSF IL-2 (pg/ml) | 8.103 (20.326)
  CSF IL-6 (pg/ml) | 21.009 (1220.991)
  CSF IL-10 (pg/ml) | -3.057 (80.133)
  CSF TNF-a (pg/ml) | -0.396 (11.426)

3. Primary Outcome: CSF Biomarkers of Pharmacodynamic Response- Cytokines
Description: Change in concentration (Average Difference) of circulating cytokines in CSF from baseline. Cytokines measured include: CSF IFN-g (pg/ml), CSF IL-1b (pg/ml), CSF IL-2 (pg/ml), CSF IL-6 (pg/ml), CSF IL-10 (pg/ml), CSF TNF-a (pg/ml).
  Mean differences (and standard deviations) from baseline values are presented for the Day 364 (end of study) sample collections for the 4 participants with complete data in the study.
Time Frame: Baseline to Day 364
Measure: Mean (Standard Deviation); unit: picogram/milliliter (pg/ml)
Arm/Group | Active BCG Immunization
Number analyzed (Participants) | 4
picogram/milliliter (pg/ml)
  CSF IFN-g (pg/ml) | -14.368 (13.773)
  CSF IL-1b (pg/ml) | 5.510 (10.867)
  CSF IL-2 (pg/ml) | -12.910 (22.841)
  CSF IL-6 (pg/ml) | 710.455 (1827.730)
  CSF IL-10 (pg/ml) | -95.078 (144.162)
  CSF TNF-a (pg/ml) | 0.300 (19.083)

4. Primary Outcome: Blood Biomarkers of AD Pathology-ATN
Description: Change in concentration (Average difference) of ATN markers of AD pathophysiology phospho-tau (217 and 181) and neurofilament light protein biomarkers in blood from baseline.
  Mean differences (and standard deviations) from baseline values are presented for the Day 364 (end of study) sample collections for the 4 participants in the study at this timepoint.
Time Frame: Baseline to Day 364
Measure: Mean (Standard Deviation); unit: picogram/milliliter (pg/ml)
Arm/Group | Active BCG Immunization
Number analyzed (Participants) | 4
picogram/milliliter (pg/ml)
  Plasma pTau217 (pg/ml) | -1.392 (5.382)
  Plasma pTau181 (pg/ml) | 0.233 (0.362)
  Plasma NfL (pg/ml) | -1.852 (5.810)

5. Primary Outcome: CSF Biomarkers of AD Pathology-ATN
Description: Change in concentration (Average difference) of ATN markers of AD pathophysiology (phospho-tau181, total tau, and neurofilament light protein biomarkers in CSF from baseline.
  Mean differences (and standard deviations) from baseline values are presented Day 364 (end of study) sample collections for the 4 participants in the study at this timepoint.
Time Frame: Baseline to Day 364
Measure: Mean (Standard Deviation); unit: picogram/milliliter (pg/ml)
Arm/Group | Active BCG Immunization
Number analyzed (Participants) | 4
picogram/milliliter (pg/ml)
  CSF tTau (pg/ml) | -3.595 (26.970)
  CSF pTau181 (pg/ml) | -5.955 (10.135)
  CSF NfL (pg/ml) | -55.413 (477.315)

6. Primary Outcome: Blood Biomarkers of AD Pathology-ATN
Description: Change in concentration (Average difference) of ATN markers of AD pathophysiology (phospho-tau (217 and 181) and neurofilament light protein biomarkers in blood from baseline.
  Mean differences (and standard deviations) from baseline values are presented for the Day 84 sample collections for the 7 participants in the study at this timepoint.
Time Frame: Baseline to Day 84
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: picogram/milliliter (pg/ml)
Arm/Group | Active BCG Immunization
Number analyzed (Participants) | 7
picogram/milliliter (pg/ml)
  Plasma pTau217 (pg/ml) | 0.916 (7.179)
  Plasma pTau181 (pg/ml) | 0.004 (1.288)
  Plasma NfL (pg/ml) | -1.735 (7.881)

7. Primary Outcome: CSF Biomarkers of AD Pathology-ATN
Description: Change in concentration (Average difference) of ATN markers of AD pathophysiology (phospho-tau181, total tau, and neurofilament light protein biomarkers in CSF from baseline.
  Mean differences (and standard deviations) from baseline values are presented for the Day 84 sample collections for the 4 participants in the study at this timepoint.
Time Frame: Baseline to Day 84
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: picogram/milliliter (pg/ml)
Arm/Group | Active BCG Immunization
Number analyzed (Participants) | 7
picogram/milliliter (pg/ml)
  CSF tTau (pg/ml) | 8.727 (49.826)
  CSF pTau181 (pg/ml) | -2.414 (11.793)
  CSF NfL (pg/ml) | -103.161 (317.523)

8. Primary Outcome: Cognitive Measures (RBANS)
Description: Change in Total Scale Index (TSI) of the Repeatable Battery for the Assessment of Neuropsychological Status (RBANS). Mean differences and standard deviations are expressed for the difference between the Day 84 TSI and the baseline TSI for the 7 participants in the study.
  The RBANS is an assessment commonly used in clinical trials to assess cognitive functioning. Scores range from 40 to 160 with lower scores indicating poorer performance, thus a score decrease would indicate a decrease in cognitive performance. A score under 78 is typically indicative of cognitive impairment.
Time Frame: Baseline to Day 84
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active BCG Immunization
Number analyzed (Participants) | 7
score on a scale | 17.710 (35.127)

9. Primary Outcome: Cognitive Measures (RBANS)
Description: Change in Total Scale Index (TSI) of the Repeatable Battery for the Assessment of Neuropsychological Status (RBANS). Mean differences and standard deviations are expressed for the difference between the end of study TSI and the baseline TSI for the 4 participants in the study.
  The RBANS is an assessment commonly used in clinical trials to assess cognitive functioning. Scores range from 40 to 160 with lower scores indicating poorer performance, thus a score decrease would indicate a decrease in cognitive performance. A score under 78 is typically indicative of cognitive impairment.
Time Frame: Baseline to Day 364
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active BCG Immunization
Number analyzed (Participants) | 4
score on a scale | -5.667 (19.075)

10. Primary Outcome: Amyloid-β42/40 Average Difference in Blood
Description: Average difference of ATN markers of AD pathophysiology (Amyloid-β42/40 ratio) in blood from baseline.
Time Frame: Baseline to Day 364
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Active BCG Immunization
Number analyzed (Participants) | 4
ratio | -0.001 (0.06)

11. Primary Outcome: Amyloid-β42/40 Average Difference in CSF
Description: Average difference of ATN markers of AD pathophysiology (Amyloid-β42/40) in CSF from baseline.
Time Frame: Baseline to Day 364
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Active BCG Immunization
Number analyzed (Participants) | 4
ratio | 0.000 (0.002)

12. Primary Outcome: Amyloid-β42/40 Average Difference in Blood - Baseline to Day 84
Description: Average difference of ATN markers of AD pathophysiology (Amyloid-β42/40) in blood from baseline.
Time Frame: Baseline to Day 84
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Active BCG Immunization
Number analyzed (Participants) | 7
ratio | 0.001 (0.005)

13. Primary Outcome: Amyloid-β42/40 Average Difference in CSF - Baseline to Day 84
Description: Average difference of ATN markers of AD pathophysiology (Amyloid-β42/40) in CSF from baseline.
Time Frame: Baseline to Day 84
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Active BCG Immunization
Number analyzed (Participants) | 7
ratio | -0.001 (0.001)

14. Primary Outcome: Blood Biomarkers of Pharmacodynamic Response - Cytokines
Description: Change in concentration of circulating cytokines in blood plasma from baseline. Cytokines include: Plasma IFN-g (pg/ml), Plasma IL-1b (pg/ml), Plasma IL-2 (pg/ml), Plasma IL-6 (pg/ml), Plasma IL-10 (pg/ml), Plasma TNF-a (pg/ml). Mean differences (and standard deviations) from baseline values are presented for the Day 84 sample collections for the 7 participants in the study at that time.
Time Frame: Baseline to Day 84
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: picograms/mililiter (pg/ml)
Arm/Group | Active BCG Immunization
Number analyzed (Participants) | 7
picograms/mililiter (pg/ml)
  Plasma IFN-g (pg/ml) | 365.612 (926.852)
  Plasma IL-1b (pg/ml) | -24.320 (100.242)
  Plasma IL-2 (pg/ml) | 0.460 (48.615)
  Plasma IL-6 (pg/ml) | -530.279 (1926.387)
  Plasma IL-10 (pg/ml) | 97.486 (269.749)
  Plasma TNF-a (pg/ml) | 12.004 (151.302)

ADVERSE EVENTS:
Time Frame: AEs were collected starting at screening through Day 364 Visit for each participant.
Arm/Group | Active BCG Immunization
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 1/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active BCG Immunization (N=15)
Elevated Blood Pressure (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-10-13): https://cdn.clinicaltrials.gov/large-docs/88/NCT05004688/Prot_SAP_000.pdf